CLINICAL TRIAL: NCT07087535
Title: Midterm Follow up Outcomes of Single Anastomosis Sleeve Jejunal Bypass (SASJ) in Management of Morbid Obesity
Brief Title: Midterm Follow up Outcomes of (SASJ) in Management of Morbid Obesity
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed Khalaf, resident, Sohag University
Other Study IDs: Soh-Med--25-6-9MS
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Morbid Obesity Requiring Bariatric Surgery
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is a critical health problem associated with an increased risk of cardiovascular disease, diabetes, and cancers, affecting both the quality of life and life expectancy . The increasing prevalence of obesity and comorbid conditions requires effective treatment and prevention . Previous evidence has demonstrated that bariatric surgery is associated with greater and longer-term weight loss than non-surgical management Thus, in patients with a body mass index of ≥ 40 or ≥ 35 kg/m2 with co-morbidities, bariatric surgery is the most effective treatment option that not only promotes weight loss but also improves comorbid conditions . However, like any surgical procedure, several complications can occur . The development of nutritional deficiencies is a complication which may be life-threatening; therefore, bariatric surgery requires careful consideration .

The most frequently performed surgery for obesity worldwide is the laparoscopic sleeve gastrectomy (LSG), the Roux-en-Y gastric bypass (RYGB), and more recently, the one anastomosis gastric bypass (OAGB) .

One newly developed weight loss procedure, the single sleeve ileal anastomosis bypass (SASI), has been developed as a modification to Santoro's operation (sleeve gastrectomy with transit bipartition SG + TB) . Since no duodenal division or manual anastomosis is required, the procedure allows easy endoscopic access to the duodenum . noted that SASI has the following advantages over other bariatric procedures: SASI has a shorter operative time compared to other procedures; 2) easy access to the duodenum and biliary tree endoscopically; 3) SASI does not divide the duodenum, thus eliminating the possibility of duodenal stump leakage, a serious complication with an incidence range between; 4) the tension on the anastomosis lower than other techniques; 5) there are no blind loops, excluded segments, or foreign bodies; 6) SASI is completely reversible .

Single anastomosis sleeve jejunal (SASJ) bypass, which is the focus of this study, is a modification of SASI using a shorter biliopancreatic limb length compared to SASI to prevent long-term nutritional complications . The SASJ bypass appears to be safer than the SASI procedure in patients with excessive weight loss and nutritional deficiencies and is simpler due to its improved surgical ergonomics .

Aim of the Work This study aims to evaluate the three-year outcomes of SASJ bypass as a primary bariatric procedure in a tertiary bariatric center for weight loss, comorbidity resolution, and both early and late complications.

DETAILED DESCRIPTION:
A retrospective study with prospective collected data included a case series of consecutive bariatric patients who underwent SASJ bypass in Sohag university hospitals between the 1st of January 2019 and the 31st of june 2023. The analysis in the present study included data of all the patients who underwent SASJ as bariatric procedure. All patients were approved as candidates for bariatric surgery by a multidisciplinary screening team, between 18 and 65 years of age and a BMI more than 40 kg/m2 or BMI of more than 35 kg/m2 combined with comorbidities.

All the required data have been collected from the patients' files at Sohag university hospitals out-patient clinic. To update follow up data for missing patients, a postal questionnaire will be sent to all patients to retrieve the latest outcome. Patients who will not respond will receive a phone call and email if applicable. The postal questionnaire contained questions about:

1. Current and lowest weight after surgery.
2. Current comorbidities and medication.
3. Possible complaints / complications.
4. Any surgical intervention related to the SASJ bypass. In case of non-response, the data of the last visit either in hospital or out-patient clinic were used as a final outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* Both sexes.
* Body mass index (BMI) > 35 with comorbidities or BMI > 40 with or without comorbidities.
* Primary bariatric procedure.
* Follow up period 2 years or more after SASJ.

Exclusion Criteria:

* Follow up period less than 2 years.
* Previous laparoscopic metabolic surgery
* Patients with huge anterior abdominal wall hernias.
* Cirrhotic patients.
* Pregnant or lactating females.
* Unfit patients for anesthesia.
* patients requiring revisional bariatric surgery.
* Patients with any contraindications to laparoscopic surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sohag University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
weight loss outcomes | 2 years
  * Percentage of excess weight loss
  * Percentage of total weight loss

SECONDARY OUTCOMES:
comorbidities readmission reoperation | 2 years
  * Comorbidity resolution
  * readmission
  * reoperation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Hospital University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT07087535/Prot_000.pdf